CLINICAL TRIAL: NCT04057209
Title: VoiceS: Voice Quality After Transoral CO2-Laser Surgery Versus Single Vocal Cord Irradiation for Unilateral Stage 0 & I Glottic Larynx Cancer - A Randomized Phase III Trial
Brief Title: VoiceS: Voice Quality After Transoral CO2-Laser Surgery Versus Single Vocal Cord Irradiation for Larynx Cancer
Acronym: VoiceS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olgun Elicin (Other)
Collaborators: University of Bern (Other); The Netherlands Cancer Institute (Other); University of Lausanne Hospitals (Other); University Hospital, Geneva (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Olgun Elicin, Principal Investigator and Sponsor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-BE 2019-01506
Record Dates: First submitted 2019-08-07; First posted 2019-08-15 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Glottis Tumor; Larynx Cancer
Keywords: head and neck cancer; squamous cell carcinoma; carcinoma in situ; radiotherapy; surgery; transoral laser microsurgery; patient reported outcome; quality of life; voice
MeSH Terms: conditions — Laryngeal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Carcinoma in Situ

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The secondary phoniatric assessments will be carried out centrally by blinded phoniatricians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Transoral CO2-Laser Microsurgical Cordectomy (TLM) (Active Comparator): Transoral CO2-Laser Microsurgical Cordectomy defined by European Laryngological Society (Remacle M, Eckel HE, Antonelli A, et al. Endoscopic cordectomy. A proposal for a classification by the Working Committee, European Laryngological Society. Eur Arch Otorhinolaryngol. 2000;257(4):227-231.)
  Interventions: Procedure: Arm A: Transoral CO2-Laser Microsurgical Cordectomy (TLM)
- Arm B: Single Vocal Cord Irradiation (SVCI) (Experimental): Single Vocal Cord Irradiation defined by Kwa et al. and Al-Mamgani et al. (Kwa SLS, Al-Mamgani A, Osman SOS, Gangsaas A, Levendag PC, Heijmen BJM. Inter- and Intrafraction Target Motion in Highly Focused Single Vocal Cord Irradiation of T1a Larynx Cancer Patients. Int J Radiat Oncol Biol Phys. 2015;93(1):190-195. Al-Mamgani A, Kwa SLS, Tans L, et al. Single Vocal Cord Irradiation: Image Guided Intensity Modulated Hypofractionated Radiation Therapy for T1a Glottic Cancer: Early Clinical Results. Int J Radiat Oncol Biol Phys. 2015;93(2):337-343.)
  Interventions: Radiation: Single Vocal Cord Irradiation (SVCI)

INTERVENTIONS:
Radiation: Single Vocal Cord Irradiation (SVCI) — The following planning aim will be pursued: full coverage of the PTV with at least 95% of the prescribed dose and a maximum (0.03 cc) PTV dose of <107%: 16 x 3.63 = 58.08 Gy in 5 fractions per week using 5 to 9 static IMRT or VMAT.
  Arms: Arm B: Single Vocal Cord Irradiation (SVCI)
Procedure: Arm A: Transoral CO2-Laser Microsurgical Cordectomy (TLM) — The TLM has to be performed using a CO2 laser, coupled to an operative microscope, at 4-8W in ultrapulse mode. The type of cordectomy performed must be mentioned using the following classification according the classification of the European Laryngological Society.
  The type of resection chosen should provide complete removal of the primary lesion with negative margins.
  Surgery will generally be performed within 3 weeks after randomization and not more than 6 weeks after panendoscopy.
  The extent of the cordectomy must include a complete anterior, posterior, inferior and supero-lateral mucosal and deep soft tissue margin.
  Arms: Arm A: Transoral CO2-Laser Microsurgical Cordectomy (TLM)

SUMMARY:
Laser surgery and radiotherapy are well-established standards of care for unilateral stage 0 & I carcinoma in situ (Cais) and squamous cell carcinoma of glottic larynx (SCCGL). Based on meta-analyses, functional and oncological outcome after both treatment modalities are comparable1-5. However, no properly conducted randomized trials comparing these treatments exist. The only such trial with the endpoint of voice quality had to be prematurely closed due to low accrual6.

The traditional radiotherapy involves the treatment of the whole larynx. Recently, a new radiotherapy technique was introduced by a team of researchers from Netherlands, where the treated target volume consists of involved vocal cord and therefore 8 to 10-fold smaller than the target volumes used for traditional whole larynx irradiation. The treatment is reduced to 16 fractions which corresponds to 3 weeks and a day7-12. The results of a prospective cohort (n=30) with single vocal cord irradiation (SVCI) were compared with the results of a historical prospective cohort previously treated with whole larynx radiotherapy (n=131) in the same institute. The median follow-up was 30 months. The voice handicap index (VHI) at all time points beginning from the 6th week after SVCI was significantly superior to the same time points with conventional radiotherapy. Moreover, a comparable local control with SVCI (100%) vs. conventional radiotherapy (92%) was reported at two years, p=0.2412.

Based on this information, the investigators' main aim is to compare SVCI to Transoral CO2-Laser Microsurgical Cordectomy (TLM) with the main focus of patient-reported voice quality.

DETAILED DESCRIPTION:
Background and Rationale

Head and neck squamous cell carcinoma (HNSCC) is the 6th most common type of cancer worldwide. Of all head and neck cancers, approximately 30% originates from the larynx. In Europe, annually 52.000 patients are diagnosed with cancer of the larynx. About 50-60% of laryngeal squamous cell carcinomas arise from the glottic region and over 80% of these patients present in an early stage. The larynx has important roles in production of voice, coordination of deglutition, and respiration. Therefore, the treatment aim of laryngeal cancer is not only achievement of maximum disease control, but also maintenance of function. Transoral CO2-Laser Microsurgical Cordectomy (TLM) and radiotherapy are well-established standard treatment modalities for unilateral stage 0-I carcinoma in situ and squamous cell carcinoma of glottic larynx (for convenience, both will be mentioned as SCCGL throughout this protocol). Based on various clinical studies and meta-analyses, functional and oncological outcome (overall survival and local control) after both treatment modalities are comparable. However, no properly conducted randomized trials comparing these treatments exist. The only such trial with the endpoint of voice quality had to be prematurely closed due to low accrual.

The treatment option varies remarkably in different countries and among institutions. Especially in the case of unilateral SCCGL, other factors such as voice quality, cultural and socioeconomic factors, and patients' preference should be considered. Hoarseness is one of the main and early signs of SCCGL, whereas both radiotherapy and TLM influence voice quality by altering the vocal cord motion and anatomy. Another issue worth to consider is the treatment time. Surgery is performed in one day followed by a few days of hospital stay. In contrast, radiotherapy is applied in daily fractions. Although each fraction only takes few minutes, the patients have to visit the radiation oncology department over a course of 4 to 7 weeks, depending on the institutional preference of dose and fractionation. The post-treatment follow-up schedules are identical for both strategies.

The differences between both treatment modalities have been extensively reported. However, either due to no meaningful difference or due to the heterogeneity in the voice analysis techniques, several studies revealed no significant differences while better voice quality was reported after radiotherapy as compared with TLM in other studies.

The traditional radiotherapy involves the treatment of the whole larynx over a period of 4 to 7 weeks. Recently, a new radiotherapy technique was introduced by a team of researchers from Netherlands, where the treated target volume consists of involved vocal cord and therefore 8 to 10 fold smaller than the target volumes used for traditional whole larynx irradiation. The treatment is reduced to 16 fractions with higher dose per fraction which corresponds to 3 weeks and a day. The results of a prospective cohort (n=30) with single vocal cord irradiation (SVCI) were compared with the results of a historical prospective cohort (n=131) previously treated with whole larynx radiotherapy in the same institute. The median follow-up was 30 months. The voice handicap index (VHI) at all time points beginning from the 6th week after SVCI was significantly superior to the same time points with conventional radiotherapy. Moreover, a comparable local control with SVCI (100%) vs. conventional radiotherapy (92%) was reported at two years, p=0.2412.

In conclusion, the long-term voice quality and oncologic outcome (survival and local tumor control) are comparable with both TLM and traditional radiotherapy. Furthermore, the new SVCI technique offers a possibly superior long-term voice quality with an at least equal oncologic outcome compared to traditional radiotherapy. With this background, the investigators' main aim is to compare SVCI to TLM with the main focus of patient-reported voice quality.

Investigational Treatments and Indication

With the indication to treat early stage SCCGL in an organ preservation setting, both TLM and SVCI are going to be compared head-to-head, and therefore are considered as investigational treatments.

Clinical Evidence to Date

In well-recognized international cancer treatment guidelines, TLM and radiotherapy are considered as comparable modalities for the successful treatment of early stage SCCGL. Based on various clinical studies and meta-analyses, functional and oncological outcome (overall survival and local control) after both treatment modalities are comparable. However, no properly conducted randomized trials comparing these treatments exist. The only such trial with the endpoint of voice quality had to be prematurely closed due to low accrual.

The differences between both treatment modalities have been extensively reported. However, either due to no meaningful difference or due to the heterogeneity in the voice analysis techniques, several studies revealed no significant differences while better voice quality was reported after radiotherapy as compared with TLM in other studies. Nevertheless, most of the literature consists of reports about retrospective case series with the lack of level I evidence.

Justification of Choice of Study Population

In line with the eligibility criteria, the study population will include patients diagnosed with unilaterally situated stage 0-I SCCGL who are considered as eligible both for radiotherapy and surgery by a multidisciplinary tumor board. Both treatment modalities are well-established standards.

Study Objectives

Overall Objective The ultimate goal of the study is to compare the treatment outcome of the SVCI and TLM for unilateral stage 0-I SCCGL.

Primary Objective Comparison of patient-reported subjective voice quality after TLM and SVCI

Secondary Objectives

* Qualitative post-therapeutic comparison of the voice between study arms
* Quantitative post-therapeutic comparison of the voice between study arms
* Comparison of the oncological outcome between study arms.
* Assessment of toxicity/morbidity among study arms with the listed toxicity items provided in Appendix A. CTCAE v.5.0 will be used for the classification of toxicities.

Safety Objectives - Assessment of toxicity/morbidity among study arms with the listed toxicity items provided in Appendix A. CTCAE v.5.0 will be used for the classification of toxicities.

Study Outcomes

Primary Outcome

- Average of the VHI assessed at 6, 12, 18, and 24 months

Secondary Outcomes

* Perceptual impression of the voice via Roughness - Breathiness - Hoarseness (RBH) assessment at 6, 12, 18, and 24 months
* Quantitative characteristics of voice by means of Jitter and Shimmer (JS), Glottal-to-Noise Excitation Ratio (GNE) and Singing Power Ratio (SPR), which will be assessed at 6, 12, 18, and 24 months
* Loco-regional control of the disease at 2 and 5 years
* Treatment toxicity at 2 and 5 years based on CTCAE v.5.0

Other Outcomes of Interest The patient, disease and procedural characteristics will be described.

Safety Outcomes Although the safety endpoints within the secondary endpoints will be published only at two time points (2 and 5 years), the toxicity will be systematically assessed during and after the treatment in a more frequent schedule: during the treatment, every 3 months until 24 months, and every 6 months between the 24th and 60th months. Assessment of toxicity/morbidity among study arms with the listed toxicity items provided in Appendix A. CTCAE v.5.0 will be used for the classification of toxicities.

Study Design

General study design and justification of design This is a prospective randomized multi-center open-label comparative phase III study with a superiority design (see Section 11 for the details of statistical considerations). Primary endpoint of this study is patient-reported subjective voice quality between 6 to 24 months after randomization.

The sample size calculation is based on the primary outcome, the VHI at 6 to 24 months (averaged). Based on the literature, the investigators consider the VHI to be comparable between TLM and traditional whole larynx radiotherapy. Therefore, the working hypothesis is that there is a difference between TLM and SVCI in regard to VHI. Al-Mamgani et al. reported standard deviations for VHI ranging from 2 to 10 score points12. A difference of 8 points between the two groups are regarded as clinically relevant and a conservative standard deviation of 8 points is assumed. Based on a two-sample means test, 34 patients (17 per group) are needed to detect a difference in VHI at a two-sided alpha-level of 0.05 with a power of 80%.

This sample size calculation is conservative. In the analysis, the average difference over four time points (6, 12, 18, and 24 months) will be modelled and additionally adjusted for the baseline VHI to yield more power. In each center, patients will be enrolled into the study by the local principal investigator. The local PI can be a head and neck surgeon or radiation oncologist. However, before patient accrual, the patient must be informed about the study at least by the attending surgeon and the radiation oncologist. It is highly recommended that the patient is evaluated and informed in a multidisciplinary tumor board setting before the accrual.

Interventions in the trial are considered as non-experimental standard treatments. No diagnostic tool or imaging modality that will be used during the trial is experimental. No interim analysis for futility or safety will be performed.

Methods of minimizing bias

Randomization A probabilistic minimization technique will be used for random treatment allocation between the two treatment arms using a 1:1 ratio. The computer chooses a treatment dynamically, based on the tumor stage (Stage 0 vs. I), and VHI at baseline (<34 vs. ≥34) as two predefined stratification factors.

Allocation will be done via a dedicated website within the clinical trial management system also containing the electronic case report forms. Only system administrators who are otherwise not involved in the trial will have access to the algorithm and stored lists during the recruitment period. Investigators receive the allocation only after registration of a patient. The underlying randomization lists and details of the minimization algorithm will not be disclosed but kept securely at CTU Bern. All these measures will help to ensure concealment of allocation.

Blinding procedures Due to obvious differences between surgery and radiotherapy, it is not possible to have a blinded design in this study setting.

ELIGIBILITY:
Inclusion Criteria

1. ECOG performance status 0-1 at the time of registration
2. ≥18 years of age
3. Baseline assessments and documentation of voice quality by means of VHI, JS, RBH, GNE, SPR
4. Histopathologically confirmed, previously untreated unilateral (cT1a or unilateral cTis) stage 0 or I glottic larynx cancer based on the UICC staging system (8th edition)
5. History and physical examination by treating physician (head and neck surgeon and radiation oncologist) within 28 days prior registration
6. The patient must be expected to withstand both study interventions
7. The patient must have undergone panendoscopy with assessment for the feasibility of transoral exposure for resection. Patients without feasible exposure are not eligible
8. Localization of the tumor should allow resection with a minimum of 2 mm macroscopical margin without extension to the contralateral vocal fold, without partial resection of the arytenoid cartilage and without resection of parts of thyroid cartilage (Cordectomy Type I-IV according the classification of the European Laryngological Society)13
9. Hemoglobin ≥10 g/dL or 6.2 mmol/L (Note: The use of transfusion to achieve Hgb ≥10 g/dL is acceptable) within the 28 days prior to accrual
10. Women with child-bearing potential and using effective contraception, and not pregnant and agree not to become pregnant (see section 8.6) during participation in the trial and 30 days after radiotherapy. A negative pregnancy test before inclusion (within 28 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and 30 days after radiotherapy.
11. Written informed consent, signed by the patient and the investigator.

Exclusion Criteria

1. Infection hampering the voice quality at the time of voice assessment
2. Involvement of the anterior commissure by the tumor
3. Previous oncologic surgery with curative intent (exception: excisional biopsies resulting in unacceptable close R0 or R1/R2 margins may be included) or radiotherapy to larynx
4. Synchronous or previous malignancies. Exceptions are adequately treated basal cell carcinoma or SCC of the skin, or in situ carcinoma of the cervix uteri, low-risk prostate cancer or breast with a cancer-free follow-up time of at least 3 years, or other previous malignancy with a progression-free interval of at least 5 years
5. Co-existing disease prejudicing survival (expected survival less than 6 months)
6. Active bacterial or fungal infection requiring intravenous antibiotics at the time of registration
7. History of any voice disorders (not related to the SCCGL) lasting longer than 3 weeks
8. Illness requiring hospitalization or precluding study therapy within 28 days before registration
9. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index | up to 2 years
  average of the VHI scores (range: 0-120) of each patient up to 24 months after randomization

SECONDARY OUTCOMES:
Roughness - Breathiness - Hoarseness (RBH) | 6, 12, 18, and 24 months
  The perceptual impression of a vocal signal remains the gold standard in phoniatric diagnosis. By means of reading the phonetically balanced text "The Rainbow Passage" in English and "Die Sonne und der Wind" in German, French and Italian (versions in different languages provided in the protocol), the speaking voice is assessed by the investigator according to the parameters roughness - breathiness - hoarseness (RBH), using the scale of 0: normal, 1: mild, 2: moderate, 3: severe. In this study, the assessment will be carried out blind.
Jitter and shimmer (JS) | 6, 12, 18, and 24 months
  JS are regarded as objective, quantitative characteristics of voice quality. They describe the variations in the fundamental note of a vocal signal. Jitter is the variation of the cycle-to-cycle frequency in held vowels (in Hz or. %, norm = 0-3%), shimmer is the cycle-to-cycle variation in the amplitude of held vowels (in dB, or. %, norm = 0-20%). In this study, the assessment will be carried out blind.
Glottal-to-Noise Excitation Ratio (GNE) | 6, 12, 18, and 24 months
  GNE serves to describe the relationship of the voice signal to the noise signal (norm = 1-0) and is also a quantitative characteristic of voice quality. Jitter, shimmer and GNE correspond to the perceptual characteristics roughness - breathiness - hoarseness. In order to carry out jitter, shimmer and GNE, the test subjects hold the vowel /a/ mezzoforte for at least 5 seconds at their average speaking pitch. The vocal samples will be recorded and subsequently evaluated using the open source freeware software Praat (http://www.fon.hum.uva.nl/praat/ by Paul Boersma and David Weenink - Phonetic Sciences, University of Amsterdam Spuistraat 210 1012VT Amsterdam, Netherlands). In this study, the assessment will be carried out blind.
Singing Power Ratio (SPR) | 6, 12, 18, and 24 months
  The 'brilliant' sound of a voice is characterized in acoustic terms by a high degree of acoustic energy above 2 kHz. This can be calculated with the aid of the SPR. In the Fast-Fourier-Transformation, the amplitudes of the highest peaks between 2 and 4 kHz and of the highest peaks between 0 and 2 kHz are determined using a vocal sample and the one subtracted from the other. The lower the SPR, the more "sonorous" is the voice. For this, the test subjects hold the vowel /a/ mezzoforte for at least 5 seconds at their average speaking pitch. The vocal samples will be recorded and subsequently evaluated using Praat. In this study, the assessment will be carried out blind.
Loco-regional control of the disease | 2 and 5 years
  Event: loco-regional failure after randomization
  The time-to-event outcome loco-regional control will be evaluated using Kaplan-Meier curves and a Cox model adjusted for the randomization stratification factors.
Toxicity / Morbidity | 2 and 5 years
  Treatment toxicity up to 5 years (based on CTCAE v.5.0) after randomization
  Treatment toxicity up to 5 years will be summarized descriptively for each group, showing the overall number of events as well as number and percentage of patients with events.
Voice Handicap Index separately assessed at 6, 12, 18, and 24 months | 6, 12, 18, and 24 months
  Voice Handicap Index separately assessed at 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Olgun Elicin, M.D., Principal Investigator — Inselspital, Bern University Hospital, 3010 Bern, Switzerland
Locations (4):
- Institut Gustave Roussy, Paris, France
- Tata Memorial Hospital Mumbai, Mumbai, Maharashtra, India
- Switzerland (2):
  - Inselspital, Bern University Hospital, Bern, Canton of Bern
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
After the finalization of the study, anonymized IPD will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the peer-reviewed publication of all primary and secondary endpoints.

REFERENCES:
- [Derived] Reinhardt P, Giger R, Seifert E, Shelan M, Riggenbach E, Terribilini D, Joosten A, Schanne DH, Aebersold DM, Manser P, Dettmer MS, Simon C, Ozsahin EM, Moeckli R, Limacher A, Caparrotti F, Nair D, Bourhis J, Broglie MA, Al-Mamgani A, Elicin O. VoiceS: voice quality after transoral CO2 laser surgery versus single vocal cord irradiation for unilateral stage 0 and I glottic larynx cancer-a randomized phase III trial. Trials. 2022 Oct 27;23(1):906. doi: 10.1186/s13063-022-06841-5. PMID 36303192